CLINICAL TRIAL: NCT06804317
Title: Effectiveness of a Supervised Multicomponent Exercise-Based Telerehabilitation Intervention on Physical Performance in Older Patients with Multiple Chronic Conditions in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Universitaria Maria Cano (Other)
Responsible Party: Principal Investigator, Catalina Lopera Muñetón, clinical professor, Fundacion Universitaria Maria Cano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 013008018-2023
Record Dates: First submitted 2025-01-15; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Non Communicable Chronic Diseases
Keywords: Exercise Therapy; elderly; telerehabilitation
MeSH Terms: conditions — Noncommunicable Diseases | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NCD´s Telerehabilitation (Experimental): 41 participants enrolled in a tele-rehabilitation program with Exercise-based interventions conducted twice weekly for three months via videoconferencing on Microsoft Teams
  Interventions: Other: telerehabilitation

INTERVENTIONS:
Other: telerehabilitation — Exercise-based interventions were conducted twice weekly for three months via videoconferencing on Microsoft Teams. The program included various components:
  Aerobic and strength training, Flexibility, Balance and coordination

SUMMARY:
Currently, the older adult population faces an increase in the prevalence of cardiopulmonary diseases, which negatively impact their quality of life by limiting their ability to perform daily activities and affecting their physical and emotional well-being. In particular, cardiovascular and respiratory diseases are among the leading causes of morbidity and mortality among older adults in Colombia. Despite advances in pharmacological treatment and medical care, physical rehabilitation remains an essential component in the management of these diseases, with physical exercise serving as one of its fundamental pillars. However, access to physical rehabilitation programs for the older adult population, particularly in rural or hard-to-reach areas, continues to pose a significant challenge. Telemedicine and Information and Communication Technologies (ICT) have emerged as viable solutions to overcome this barrier, enabling the remote prescription and monitoring of physical exercises, facilitating the inclusion of more patients in rehabilitation programs, and improving their quality of life. Therefore, this study aims to evaluate the effectiveness of a multicomponent ICT-mediated intervention in terms of improving physical condition, reducing frailty, adherence, satisfaction, and quality of life in older adults with cardiopulmonary diseases.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of a non-communicable disease.
* Ability to communicate verbally or in writing.
* Stable disease status confirmed by clinical history.
* Condition present for at least three months to qualify as chronic.
* For patients with type II diabetes mellitus: glucose levels below 200 mg/dL during tele-rehabilitation sessions.

Exclusion Criteria

* Requirement for assistance with walking.
* History of disease exacerbation within the past six months.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline and at 1 month postest
  This battery includes tests for usual walking speed over 4 meters, five-chair stands, and balance. Each task receives a score (0-4) based on the time required to perform five sit-to-stand repetitions, standing balance, and walking speed over 4 meters. The total score (0-12) is calculated by summing individual scores, with higher scores indicating better lower-body function.

SECONDARY OUTCOMES:
Six-minute walk test | Baseline and at 1 month postest
  Conducted on a straight, level, hard surface, ideally 30 meters long, with a minimum acceptable length of 20 meters. The track was marked every 3 meters, with cones at the ends and bright tape at the start. Variables recorded included meters (m), which represent the total distance covered by the individual during the six-minute period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación universitaria María Cano, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No